CLINICAL TRIAL: NCT04831528
Title: The Role of Circulating Tumor DNA in Decision-making of Patients With Metastatic Colorectal Cancer After Failure of First-line Treatment Containing Cetuximab - a Single-center, Phase II Clinical Study
Brief Title: Decision-making of ctDNA in Patients With mCRC After Failure of First-line Treatment Containing Cetuximab - a Single-center, Phase II Clinical Study
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: FDZL-ctDNA
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- No secondary changes of drug resistance
  Interventions: Drug: Cetuximab Ab; Bevacizumab; Vermofenib + cetuximab;Trastuzumab+lapatinib or trastuzumab+pertuzumab; others
- Secondary mutations of RAS
  Interventions: Drug: Cetuximab Ab; Bevacizumab; Vermofenib + cetuximab;Trastuzumab+lapatinib or trastuzumab+pertuzumab; others
- Secondary mutation of BRAF
  Interventions: Drug: Cetuximab Ab; Bevacizumab; Vermofenib + cetuximab;Trastuzumab+lapatinib or trastuzumab+pertuzumab; others
- HER2 amplification
  Interventions: Drug: Cetuximab Ab; Bevacizumab; Vermofenib + cetuximab;Trastuzumab+lapatinib or trastuzumab+pertuzumab; others
- Other secondary mutations
  Interventions: Drug: Cetuximab Ab; Bevacizumab; Vermofenib + cetuximab;Trastuzumab+lapatinib or trastuzumab+pertuzumab; others

INTERVENTIONS:
Drug: Cetuximab Ab; Bevacizumab; Vermofenib + cetuximab;Trastuzumab+lapatinib or trastuzumab+pertuzumab; others — After PD, patients received ctDNA testing, and different research protocols were selected according to different gene states of ctDNA, as follows: 1.No secondary changes related to drug resistance were found. Cetuximab cross-line + second-line chemotherapy (FOLFOX/FOLFIRI/ Irinotecan monotherapy, etc.) was used.2. If there is a RAS secondary mutation, change of beacizumab bead sheet resistance + second-line chemotherapy (FOLFOX/XELOX/stand for kang single-agent FOLFIRI mXEIRI/Iraq, etc.);3. If BRAF secondary mutation occurs, replace it with vimofenib + cetuximab + irinotecan;4. If HER2 amplification occurs, replace it with trastuzumab + lapatinib or trastuzumab + pertuzumab;5. In case of other secondary mutations, bevacizumab plus second-line chemotherapy should be replaced.

SUMMARY:
This study aimis at detecting the genomic changes of ctDNA in patients of RAS and BRAF wild-type mCRC, who failed after first line treatment containing cetuximab. According to the results of ctDNA detection, individualized second-line targeted therapy strategies were developed to explore the disease control rate and prognostic significance of ctDNA-guided treatment for metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, gender unlimited;
2. Proven histologically by colorectal adenocarcinoma, local lesions can not be radical resection or metastatic colorectal cancer;
3. Patients with RAS and BRAF wild-type tissue genetic testing, receiving first-line treatment containing cetuximab, and radiographic evaluation of disease progression;
4. Eastern Cooperative Oncology Group (ECOG) physical condition score (PS) 0 ~ 2;
5. Expected survival of more than 3 months;
6. Within 7 days before screening (including 7 days), laboratory test data requirements were as follows: neutrophil count ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90g/L (no blood transfusion within 14 days), serum total bilirubin ≤1.25 times the upper normal limit (ULN);ALT and AST≤ 2.5 x ULN (≤5x ULN in patients with liver metastasis);Serum creatinine ≤1.0 x ULN and creatinine clearance rate ≥60 mL /min;Left ventricular ejection fraction in ultrasound examination >55%;
7. At least one measurable lesion (RECIST 1.1 criteria);
8. Subjects (or their legal representative/guardian) must sign the informed consent indicating that they understand the purpose of the study, understand the necessary procedures of the study, and are willing to participate in the study.

Exclusion Criteria:

Those who have one or more of the following will not be included in the study:

1. Have received any experimental drugs or anti-tumor drugs within 4 weeks before enrollment;
2. A history of other tumors in the past five years, except for cervix cancer or basal cell carcinoma of the skin that has been cured;
3. Patients with obvious intracranial hypertension or neuropsychiatric symptoms due to uncontrolled primary brain tumor or central nerve metastatic tumor
4. Pregnant or lactating women;Those who are fertile but do not take adequate contraceptive measures;
5. Alcoholism or drug addiction;
6. with pleural effusion or ascites, causing respiratory syndrome (≥CTCAE2 grade dyspnea), requiring local treatment;
7. Patients with the following serious or uncontrolled diseases: severe heart disease, unstable condition after treatment, myocardial infarction, congestive heart failure, unstable angina pectoris, pericardial effusion with obvious symptoms or unstable arrhythmia within 6 months before enrollment;Definite neuropathy or psychosis, including dementia or seizures;Severe or uncontrolled infections;Patients with active and disseminated intravascular coagulation and significant bleeding tendency
8. known hypersensitivity or anaphylaxis to any component of the study drug to be applied.
9. The function of important organs is obviously impaired
10. Other circumstances under which the investigator considers that the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ≥18y
Study Population: Patients who met the entry criteria, failed after receiving first-line treatment containing cetuximab, and were judged to have progressive disease (PD) by imaging evaluation were eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-10 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | April 10,2021-June 30,2021
  The percentage of patients whose tumors shrink by a certain amount and remain so for a certain amount of time, including patients with CR and PR.Objective tumor response was assessed using the Response Assessment Criterion for Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
overall survival | April 10,2021-June 30,2021
  Time from enrollment to death from any cause.Lost visitors to the last follow-up time.
progress free survival | April 10,2021-June 30,2021
  Patients were randomized to solstice for any recorded time of tumor progression or death from any cause.
Safety and tolerability | April 10,2021-June 30,2021
  NCI -- CTC AE 4.0 will be used to evaluate the clinical safety of the treatment in the study.The incidence of adverse events in the subjects should be assessed at each clinical visit.
duration of response | April 10,2021-June 30,2021
  This is the time between the first assessment of a tumor as CR or PR and the first assessment as PD or death from any cause.